CLINICAL TRIAL: NCT06870955
Title: Research on the Development and Clinical Evaluation of Biomimetic Abutments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stomatological Hospital Affiliated with Fujian Medical University (Other)
Responsible Party: Principal Investigator, Cheng Hui, Professor of Prosthodontics, Stomatological Hospital Affiliated with Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20211212
Record Dates: First submitted 2025-03-01; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- biomimetic abutment group (Experimental): The biomimetic healing abutments were placed during the second-stage surgery, and the biomimetic prosthetic abutments were used to complete the implant restoration.
  Historical or external data from other sources were used as controls to evaluate the treatment efficacy in the experimental group.
  Interventions: Procedure: using biomimetic abutments

INTERVENTIONS:
Procedure: using biomimetic abutments — The subjects recieved the biomimetic healing abutments during the second-stage surgery, and the biomimetic prosthetic abutments were used to complete the implant restoration.

SUMMARY:
This study aims to evaluate the clinical effectiveness of biomimetic abutments in implant restoration.

DETAILED DESCRIPTION:
The biomimetic healing abutments were placed during the second-stage surgery, and the biomimetic prosthetic abutments were used to complete the implant restoration.

To assess soft tissues, digital models were collected in STL files at five time points: before the second-stage surgery, before the implant impression, immediately after restoration, six months after restoration, and 12 months after restoration. These models were analyzed using 3D software for model matching and measurement based on CBCT, focusing on the changes on soft tissue height, width, and volume.

Hard tissue evaluation was conducted through periapical radiographs taken at three time points: immediately after restoration, six months after restoration, and 12 months after restoration.

Additionally, general clinical conditions were assessed at the same three time points, evaluating parameters such as food impaction, plaque index, and gingival index.

ELIGIBILITY:
Inclusion Criteria:

* aged between 25 and 65 years old
* had one single edentulous site
* implant embedded healed and required secondary surgery to expose
* good treatment compliance and could attend follow-up appointment regularly

Exclusion Criteria:

* soft tissue grafting was needed
* severe acute or chronic periodontitis
* heavy smoking habit (> 10 cigarettes/day)
* poor oral hygiene

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in soft tissue contour | before the second-stage surgery, before the implant impression, immediately after restoration, six months after restoration, and 12 months after restoration
  Changes of soft tissue contour in height, width, and volume by matching digital models at different treatment stages.

SECONDARY OUTCOMES:
Changes in hard tissue contour | immediately after restoration, six months after restoration, and 12 months after restoration
  Changes of hard tissue contour in height through periapical radiographs using a long-cone paralleling technique with a film holder.
Food impaction | immediately after restoration, six months after restoration, and 12 months after restoration
  Incidence of food impaction： Dichotomous registration, 0 = Absent; 1 = Present.
Plaque index | immediately after restoration, six months after restoration, and 12 months after restoration
  0 = No plaque at the gingival margin; 1 = Thin plaque layer on the gingival margin, not easily visible on inspection but detectable by scraping with a probe; 2 = Moderate plaque accumulation at the gingival margin or interproximal surfaces; 3 = Heavy plaque accumulation in the gingival sulcus, at the gingival margin, or on interproximal surfaces. Mean values among the 6 sites were obtained (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual and disto-lingual).
Gingival index | immediately after restoration, six months after restoration, and 12 months after restoration
  0 = Normal gingiva; 1 = Slight gingival edema, no bleeding on probing; 2 = Gingival edema with bleeding on probing; 3 =Tendency for spontaneous bleeding or presence of ulceration. Mean values among the 6 sites were obtained (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual and disto-lingual).

CONTACTS AND LOCATIONS:
Overall Officials: Hui Cheng, PhD, Principal Investigator — Stomatological Hospital Affiliated with Fujian Medical University
Locations (1):
- The Affiliated Stomatological Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No